CLINICAL TRIAL: NCT07068178
Title: Evaluating the Efficacy of Hyperthermic Intraperitoneal Treatment to Enhance the Sensitivity of Immune Checkpoint Inhibitor in Patients With Advanced Ovarian Cancer： A Single-arm Study
Acronym: ICI-HIPET
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jing Li (Other)
Responsible Party: Sponsor-Investigator, Jing Li, Chief Physician, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Organization: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICI-HIPET
Record Dates: First submitted 2025-06-13; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: HIPEC; Ovarian Serous Adenocarcinoma
Keywords: ICI-HIPET

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICI-HIPET (Experimental): Patients received the following interventions: On Day 0, intravenous administration of tislelizumab (an anti-PD-1 immune checkpoint inhibitor) was initiated within 3 hours post-HIPEC. Tumor tissue samples were collected before HIPEC, at 30 minutes, 60 minutes, and 90 minutes (end of HIPEC). Serum samples were collected pre- and post-HIPEC. On Day 1, additional serum samples were collected 24 hours after HIPEC-ICI completion. From Days 2-3, patients underwent paclitaxel + carboplatin chemotherapy, with serum sampling repeated at 48 hours post-HIPEC-ICI. On Days 21 and 42, the second and third cycles of neoadjuvant chemotherapy (tislelizumab + paclitaxel + carboplatin) were administered intravenously.
  Interventions: Drug: ICI-HIPET

INTERVENTIONS:
Drug: ICI-HIPET — Patients received the following interventions: On Day 0, intravenous administration of tislelizumab (an anti-PD-1 immune checkpoint inhibitor) was initiated within 3 hours post-HIPEC. Tumor tissue samples were collected before HIPEC, at 30 minutes, 60 minutes, and 90 minutes (end of HIPEC). Serum samples were collected pre- and post-HIPEC. On Day 1, additional serum samples were collected 24 hours after HIPEC-ICI completion. From Days 2-3, patients underwent paclitaxel + carboplatin chemotherapy, with serum sampling repeated at 48 hours post-HIPEC-ICI. On Days 21 and 42, the second and third cycles of neoadjuvant chemotherapy (tislelizumab + paclitaxel + carboplatin) were administered intravenously.

SUMMARY:
Background:

Advanced ovarian cancer is a highly dangerous disease, and many patients lose their lives due to limited treatment effectiveness. Previous studies have shown that current immunotherapy (e.g., PD-1 inhibitors) has poor results in ovarian cancer. The research team discovered that adding "heated abdominal chemotherapy" (called HIPEC, which uses a heated drug solution to wash the abdomen) to standard chemotherapy helps patients better control tumors. Recent lab studies also found that HIPEC not only reduces "harmful cells" around tumors that block drug effectiveness but also makes immunotherapy drugs work better. Animal experiments further confirmed that combining HIPEC with immunotherapy improves outcomes. Therefore, the investigators aim to test a key question: Can HIPEC help immunotherapy drugs work more effectively in humans?

Study Details:

The study will conduct a small two-phase trial, planning to enroll 30 patients with advanced ovarian cancer (Stage IIIc-IVA). All participants will receive standard chemotherapy (paclitaxel + platinum drugs) combined with HIPEC and an immunotherapy drug (tislelizumab, a PD-1 inhibitor). The main goal is to check whether tumors are completely removed after surgery. Investigators will also track how long tumors stay under control, overall survival time, treatment safety, and use blood and tumor tissue tests to find biomarkers that predict treatment response.

Why This Matters:

The study hopes to identify a safe method to enhance immunotherapy effectiveness and offer improved outcomes for advanced ovarian cancer patients.

DETAILED DESCRIPTION:
Advanced ovarian cancer carries a high mortality rate, and improving prognosis remains a clinical challenge, particularly given the limited efficacy of immunotherapy observed in prior studies. Prior randomized controlled trial demonstrated that hyperthermic intraperitoneal chemotherapy (HIPEC) enhances the effects of neoadjuvant chemotherapy in ovarian cancer. Further preclinical studies revealed that HIPEC reduces cancer-associated fibroblasts (CAFs) in the tumor microenvironment, alleviates immunosuppressive phenotypes, and synergizes with immune checkpoint inhibitors (ICIs) in animal models. Building on this evidence, it is hypothesized that HIPEC sensitizes ovarian cancer to ICIs. This prospective single-arm trial employs a Simon's two-stage design to evaluate HIPEC combined with tislelizumab (an anti-PD-1 agent) and standard neoadjuvant chemotherapy (paclitaxel/platinum) in 30 patients with FIGO stage IIIc-IVA high-grade serous ovarian cancer. The primary endpoint is R0 resection rate, with secondary endpoints including progression-free survival, overall survival, safety, pathological response, and multi-omics biomarker exploration. The study aims to validate HIPEC's role in enhancing ICI efficacy and provide evidence for improving immunotherapy outcomes in advanced ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with FIGO stage IIIC-IVA high-grade serous ovarian adenocarcinoma (histologically confirmed).
* Aged 18-70 years.
* Life expectancy ≥12 months.
* CT Suidan score ≥7 and Fagotti score ≥8 (assessed by two independent gynecologic oncologists via laparoscopic evaluation).
* Adequate organ function:AST/ALT ≤2× upper limit of normal (ULN);Total bilirubin ≤1.5× ULN;Serum creatinine ≤1.5× ULN.
* No myelosuppression:Hemoglobin (Hb) ≥80 g/L,White blood cell count (WBC) ≥2.0×10⁹/L,Neutrophil count ≥1.0×10⁹/L,Platelet count ≥100×10⁹/L.
* Performance Status (PS) score 0-1.

Exclusion Criteria:(Excluded if any criterion is met)

* Partial or complete bowel obstruction.
* Intestinal fistula of any grade.
* Hydronephrosis unrelieved by ureteral stenting.
* History of organ transplantation.
* Inflammatory bowel disease.
* Active or history of autoimmune diseases (e.g., systemic lupus erythematosus).
* Prior immunotherapy (including cellular therapy) or use of immunomodulators.
* Brain metastases.
* Grade ≥3 venous thromboembolism.
* Active infections (e.g., tuberculosis).
* Prior pelvic/abdominal radiotherapy.
* Prior hyperthermic intraperitoneal chemotherapy (HIPEC) or thermotherapy.
* Grade ≥2 dysfunction of major organs (e.g., heart, liver, kidneys).
* Other malignancies within 5 years (except skin or thyroid cancer).
* Psychiatric disorders affecting compliance.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
R0 Resection Rate | At interval debulking surgery (approximately 9-12 weeks after treatment initiation)
  R0 resection rate refers to the proportion of patients achieving complete macroscopic tumor removal (no visible residual disease) during interval debulking surgery after three cycles of neoadjuvant chemotherapy. This is determined by the surgeon's intraoperative assessment of the pelvic and abdominal cavities for any gross residual lesions.

SECONDARY OUTCOMES:
Rate of progression-free survival | From day 1 of treatment until progression/death, through study completion (up to 24months)
  The 1-year, 2-year, and median progression-free survival (PFS) rates of patients were calculated.
Rate of overall survival | From completion of first neoadjuvant therapy until death from any cause, assessed up to 24 months
  The 1-year, 2-year overall survival (OS) rates and median OS of patients were calculated.
Pathological response rate | During pathological examination of omental tissue (within 2 weeks post-surgery)
  Independently assessed by pathologists, defined as the absence of microscopic residual tumor in all specimens obtained during interval debulking surgery.
  Incidence of chemotherapy response score 3 (CRS3): Following three cycles of neoadjuvant therapy, patients underwent surgical debulking via laparotomy. The omental tissue was evaluated using the chemotherapy response score (CRS) system to determine the rate of CRS3 (indicating complete or near-complete pathological response).
Radiological Response Rate | After 3 cycles of neoadjuvant therapy (approximately 9 weeks)
  Independently assessed by radiologists using baseline CT or MRI (prior to neoadjuvant therapy) as reference. Tumor changes were evaluated after three cycles of neoadjuvant therapy, categorized as follows:
  Complete Response (CR): Disappearance of all target lesions, except for nodal disease. All target nodes must shrink to normal size (short axis <10 mm). All lesions must be assessed.
  Partial Response (PR): ≥30% reduction in the sum of diameters of all measurable target lesions compared to baseline. Nodal lesions are measured by short axis, while non-nodal lesions use the longest diameter. All lesions must be assessed.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters relative to the smallest value recorded during the study (or baseline if no decrease was observed), plus an absolute increase of ≥5 mm. Appearance of new lesions also qualifies as PD.
  Stable Disease (SD): Neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD

OTHER OUTCOMES:
Adverse Event (AE) Incidence | up to 24 months
  Adverse events occurring during the study were evaluated and recorded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0. Data included the number of patients (incidence), type of events, and severity (graded from Grade 1 to Grade 5 based on CTCAE criteria).

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Don't share IPD